CLINICAL TRIAL: NCT03511885
Title: EUROASPIRE V Survey on Cardiovascular Disease Prevention and Diabetes
Acronym: EUROASPIRE
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: European Society of Cardiology (Network)
Responsible Party: Sponsor
Other Study IDs: 16HH3189
Record Dates: First submitted 2018-04-16; First posted 2018-04-30 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Cardiovascular Diseases; Coronary Heart Disease
Keywords: Cardiovascular; Prevention; EUROASPIRE
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples for measuring lipids, glucose, HbA1c and creatinine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- high cardiovascular risk patients: Coronary patients
  * Elective coronary artery bypass surgery (CABG).
  * Elective percutaneous coronary intervention (PCI) .
  * Acute coronary syndromes (acute myocardial infarction with ST elevation (STEMI) and Non ST elevation MI (Non- STEMI) including those treated with primary PCI and/or CABG, and unstable angina).
  People at high risk of cardiovascular disease (CVD) who have been prescribed one or more of the following medications: (i) blood pressure and/or (ii) lipid and/or (iii) glucose lowering (diet and/or oral hypoglycaemic agents and/or insulin) treatments prescribed by a physician.
  Interventions: Other: There is no intervention

INTERVENTIONS:
Other: There is no intervention

SUMMARY:
EUROASPIRE is a multicentre European study in coronary patients and individuals at high risk of developing cardiovascular disease (CVD), describing their management through lifestyle and use of drug therapies and providing an objective assessment of clinical implementation of current scientific knowledge. Four EUROASPIRE surveys have been carried out by the European Society of Cardiology so far: EUROASPIRE I in 1995-1997 in nine countries, EUROASPIRE II in 1999- 2000 in 15 countries, EUROASPIRE III in 2006-2009 in 22 countries and EUROASPIRE IV in 2012-2015 in 26 countries. The results showed a wide gap between the recommendations and clinical practice with many patients not achieving the lifestyle and medical risk factors goals for CVD prevention. The fifth EUROASPIRE survey is planned for 2016-2018 to determine in hospital coronary patients and apparently healthy individuals in primary care at high risk of developing cardiovascular disease whether the European and national guidelines on cardiovascular disease prevention have been followed and if the practice of preventive cardiology in EUROASPIRE IV has improved by comparison with those centres which took part in EUROASPIRE I, II, III and IV. This survey will also incorporate an assessment of dysglycaemia and kidney function in all patients. The main outcome measures will be the proportions of coronary and high cardiovascular risk patients achieving the lifestyle, risk factor and therapeutic targets for cardiovascular disease prevention. The data collection will be based on a review of patient medical records and a patient interview and examination at least 6 months and at most 3 years after recruiting event. All countries which participated in the first three surveys will be invited to take part in EUROASPIRE V. This fifth survey will give a unique picture of preventive action by cardiologists and primary care physicians looking after patients with coronary disease and individuals at high CVD risk.

DETAILED DESCRIPTION:
A fifth European survey of Cardiovascular Disease prevention and Diabetes (EUROASPIRE V) is being conducted in 2016-2018 under the auspices of the European Society of Cardiology, EURObservational Research Programme. This fifth survey incorporate an assessment of dysglycaemia and kidney function in all patients. As in the previous EUROASPIRE surveys this survey focusses on hospital patients with coronary heart disease, with and without diabetes mellitus, and apparently healthy individuals in primary care at high risk of developing cardiovascular disease including those with diabetes.

This multicentre European study identifies risk factors in coronary patients and high-risk individuals, describes their management through lifestyle and use of drug therapies providing an objective assessment of clinical implementation of scientific knowledge as reflected in current European management guidelines. For the first time we extended this new survey to include more information about medication adherence, atrial fibrillation, familial hypercholesterolemia and statin intolerance as risk factors for cardiovascular disease. All centres and countries that participated in the first four surveys are invited to participate in the fifth European Survey of Cardiovascular Disease Prevention and Diabetes (EUROASPIRE V) and new countries and centres will be included. This fifth survey will give a unique European picture of preventive action by cardiologists, other specialists and primary care physicians looking after patients with coronary disease and their families, individuals at high risk of developing CVD and all those with dysglycaemia, diabetes and chronic kidney disease (CKD) in Europe.

ELIGIBILITY:
Inclusion Criteria:

I. Coronary patients

Patients may fulfil more than one of the following diagnostic criteria:

i. Elective CABG. ii. Elective PCI . iii. Acute coronary syndromes (acute myocardial infarction with ST elevation (STEMI) and Non ST elevation MI (Non-STEMI) including those treated with primary PCI and/or CABG, and unstable angina).

II. High risk individuals

Three diagnostic groups will be identified by their drug treatment:

i. Antihypertensive drugs and/or ii. Lipid lowering drugs and/or iii. Glucose lowering treatments (diet and/or oral hypoglycaemics and/or insulin) Patients identified by each of these drug treatments may also be taking one or more of the other drug therapies.

Exclusion Criteria:

I. Coronary patients i. Age > 80 years ii. Severe physical disability iii. Impaired cognitive function iv. Patients admitted to hospital from outside the geographical area

II . High Risk Individuals i. History of coronary heart disease ii. Age > 80 years iii. Severe physical disability iv. Impaired cognitive function

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: I. Participating countries Belgium, Bosnia&Hertzegovina, Bulgaria, Croatia, Cyprus, Czech Republic, Egypt, Finland, France, Germany, Greece, Hungary, Ireland, Kazakhstan, Kyrgyzstan, Latvia, Lithuania, the Netherlands, Poland, Portugal, Romania, Russia, Serbia, Sweden, Slovenia, Spain, Turkey, Ukraine and the UK.
Sampling Method: Non-Probability Sample
Enrollment: 1736 (Actual)
Dates: Start 2016-08-23 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
Proportions of hospital coronary patients and high risk individuals in primary care achieving European lifestyle, risk factors and therapeutic targets for cardiovascular disease prevention | 29 months
  The management of risk in terms of lifestyle intervention and the use of drug therapies will be evaluated in relation to the lifestyle and therapeutic goals defined in the national and European guidelines on cardiovascular disease prevention.
  smoking prevalence BMI in kg/m2 blood pressure in mmHg Total cholesterol in mmol/L LDL-cholesterol in mmol/L HDL-cholesterol in mmol/L glucose in mmol/L HbA1c in %
  cardioprotective medication by drug class

CONTACTS AND LOCATIONS:
Overall Officials: David Wood, PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No